CLINICAL TRIAL: NCT04600583
Title: A Prospective, Randomized, Controlled Trial of Mechanical Axis With Soft Tissue Release Balancing vs Functional Alignment With Bony Release Balancing in Total Knee Replacement - A Study Using Stryker Mako Robotic-Arm Assisted Technology®.
Brief Title: A Trial of Mechanical Axis With Soft Tissue Release Balancing vs Functional Alignment With Bony Release Balancing in Total Knee Replacement Using Stryker's Mako Robot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker South Pacific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAMELOT
Record Dates: First submitted 2020-09-29; First posted 2020-10-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis
Keywords: Knee; Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Alignment according to Functional Alignment philosophy (Active Comparator): Patients randomized to this group will undergo a TKA (total knee arthroplasty) to receive a Triathlon Total Knee System aligned according to Functional Alignment philosophy. This method of implant alignment is defined by a patient's native joint line as well as the soft tissue envelope. Triathlon Total Knee System components will be positioned relative to intra-operative soft tissue laxity assessment. A mobile application (KneeBalancer) will be used to assist surgeon decision making during the dynamic joint balancing surgical step.
  Interventions: Device: Triathlon® Total Knee System (Stryker Orthopaedics, Mahwah, NJ USA)
- Alignment to the patient's natural Mechanical axis (Active Comparator): Patients randomized to this group will undergo a TKA (total knee arthroplasty) to receive a Triathlon Total Knee System neutrally aligned to the Mechanical axis. More specifically, the femoral component and tibial component are aligned 0° to the mechanical axis of each respective limb. Femoral component rotation is fixed to the trans-epicondylar axis. Soft tissue releases are performed at the discretion of the surgeon to achieve balance and full range of motion.
  Interventions: Device: Triathlon® Total Knee System (Stryker Orthopaedics, Mahwah, NJ USA)

INTERVENTIONS:
Device: Triathlon® Total Knee System (Stryker Orthopaedics, Mahwah, NJ USA) — All patients, regardless of the alignment arm they are randomized to will undergo a primary total knee arthroplasty with the Triathlon® Total Knee System using Mako Robotic-Arm Assisted Technology. The surgical intervention will be administered by a physician wherein the expected duration of surgery is approximately 1.5 hours.

SUMMARY:
This study is a prospective, randomized, longitudinal study of the clinical outcomes of osteoarthritis patients treated by two different alignment philosophies for total knee replacement. All patients will be treated with the same knee system, implanted using MAKO robotic-arm assisted technology.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female between the ages of 40-80 years.
* The patient requires a primary total knee replacement and is indicated for robotic-assisted surgery.
* Patient is deemed appropriate for a cruciate retaining knee replacement.
* The patient has a primary diagnosis of osteoarthritis (OA).
* The patient has intact collateral ligaments.
* The patient is able to undergo CT scanning of the affected limb.
* The patient has signed the study specific, ethics-approved, Informed Consent document.
* The patient is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations.

Exclusion Criteria:

* The patient has a history of total, unicompartmental reconstruction or fusion of the affected joint.
* Patient has had a previous osteotomy around the knee.
* The patient is morbidly obese (BMI ≥ 40).
* The patient has a deformity which will require the use of stems, wedges or augments in conjunction with the Triathlon Total Knee System.
* The patient has a varus/valgus deformity ≥ 15°.
* The patient has a fixed flexion deformity ≥ 15°.
* The patient has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
* The patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
* Patient has a cognitive impairment, an intellectual disability or a mental illness.
* The patient is pregnant.
* The patient has metal hardware present in the region of the hip, knee or ankle (as this is known to create geometrical distortion in the region of the implant).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Joint feeling and Forgotten Joint Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months (primary timepoint) and 24 months
  To evaluate differences in joint feeling assessed via the Forgotten Joint Score. This newly-developed 12-item score ranges from 0 to 100 and assesses how aware recipients are of their joint in everyday life. Higher scores indicate a good outcome i.e. a high degree of forgetting the joint. For the purpose of this study a change in score of 14 points for the Forgotten Joint Score has been identified.

SECONDARY OUTCOMES:
Function and Oxford Knee Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Oxford Knee Score. This score ranges from 0 to 48 where a higher score indicates a better outcome.
Function and The International Knee Society Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 12 months and 24 months
  To evaluate differences in function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: The International Knee Society Score. This score ranges from 0 to 100 where a higher score correlates to a better outcome.
Function and Knee Injury and Osteoarthritis Outcome Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Knee Injury and Osteoarthritis Outcome Score. This score ranges from 0 to 100 where 0 indicates the worst possible knee symptoms and 100 signifies no knee symptoms.
Pain and Oxford Knee Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in pain between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Oxford Knee Score. This score ranges from 0 to 48 where a higher score indicates a better outcome.
Pain and The International Knee Society Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 12 months and 24 months
  To evaluate differences in pain between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: The International Knee Society Score. This score ranges from 0 to 100 where a higher score correlates to a better outcome.
Pain and Knee Injury and Osteoarthritis Outcome Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in pain between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Knee Injury and Osteoarthritis Outcome Score. This score ranges from 0 to 100 where 0 indicates the worst possible knee symptoms and 100 signifies no knee symptoms.
Pain and Visual Analogue Scale | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in pain between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following graphic measurement instrument: Visual Analogue Scale. This scale is a continuum between no pain and the worst possible pain imaginable.
Satisfaction and Net Promoter Score | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in satisfaction between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Net Promoter. This score ranges from -100 to 100 where the upper end indicates the patient's recommendation of the healthcare they received.
Health related quality of life and Euro-Qol (EQ-5D-3L) | Pre-operative (2 weeks prior to surgery), Post-operative - 6 weeks, 6 months, 12 months and 24 months
  To evaluate differences in health-related quality of life between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This will be achieved by employing the following instrument: Euro-Qol (EQ-5D-3L). This score ranges from 0 to 100 where 0 correlates to the worst imaginable health state whilst 100 indicates the best.
Early pain | In-patient setting (< 5 days post-operation), Post-operative - 6 weeks and 6 months
  To evaluate differences in early pain (i.e. from in-patient setting to 6-months post operation) between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved through the use of a patient pain inventory form.
Early function | In-patient setting (< 5 days post-operation)
  To evaluate differences in early function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved by utilizing functional tests conducted by physiotherapists. The following functional test will be carried out on the knee joint: Range of motion
Early function | In-patient setting (< 5 days post-operation)
  To evaluate differences in early function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved by utilizing functional tests conducted by physiotherapists. The following functional test will be employed: 9 step stair climb
Early function | In-patient setting (< 5 days post-operation)
  To evaluate differences in early function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved by utilizing functional tests conducted by physiotherapists. The following functional test will be employed: fast paced 10m walk test
Early function | In-patient setting (< 5 days post-operation)
  To evaluate differences in early function between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved by utilizing functional tests conducted by physiotherapists. The following functional test will be employed: 30 second chair stand test
Blood loss | Intra-operative
  To compare blood loss between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved through obtaining surgical data.
Adjustments to balance | Intra-operative
  To compare adjustments to balance between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This objective will be achieved through obtaining the position from the Robotic system.
Ability to reach target knee balance as assessed by alignment angles and gaps | Pre-operative (2 weeks prior to surgery), intra-operative, Post-operative - 6 weeks, 12 months and 24 months
  To compare the ability to achieve soft tissue balance between Robotic Assisted Functional Alignment and Robotic Assisted Mechanical Alignment. This object will be achieved by comparing pre-operative plan and pre-resection gaps with the final surgical plan and implanted gaps as derived from the robotic system. The implant position is defined as the angulation of components and resected bone in each anatomical plane. The soft tissue balance is defined as gaps created in extension and 90° of flexion when stressing the medial compartment (medial collateral ligament) and lateral compartment (lateral collateral ligament). The overall limb alignment is assessed by comparing the Hip-Knee-Ankle angle from pre-operative to 1-year post-operative on a long leg weight bearing x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Young, Dr, Principal Investigator — North Shore Hospital
Locations (1):
- North Shore Hospital, Takapuna, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young SW, Zeng N, Tay ML, Fulker D, Esposito C, Carter M, Bayan A, Farrington B, Van Rooyen R, Walker M. A prospective randomised controlled trial of mechanical axis with soft tissue release balancing vs functional alignment with bony resection balancing in total knee replacement-a study using Stryker Mako robotic arm-assisted technology. Trials. 2022 Jul 20;23(1):580. doi: 10.1186/s13063-022-06494-4. PMID 35858944